CLINICAL TRIAL: NCT04418635
Title: Herbal Supplement Prosta-OK® Neo as an Adjunct Therapy in Patients With Mild to Severe Non-neurogenic Male Lower Urinary Tract Symptoms Receiving Tamsulosin Therapy: a Double-blind, Randomized, Placebo-controlled Trial.
Brief Title: Herbal Supplement Prosta-OK® Neo as an Adjunct Therapy in Patients With Mild to Severe Non-neurogenic Male Lower Urinary Tract Symptoms Receiving Tamsulosin Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acrobio Healthcare Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: LPO201910
Record Dates: First submitted 2020-05-18; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-05

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: lower urinary tract symptoms; International Prostate Symptom Score; tamsulosin; adjunct therapy; herbal extractions; double-blind; randomized controlled trial
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tamsulosin and Prosta-OK® Neo (Experimental): Tamsulosin 0.2mg once daily and Prosta-OK® Neo 707mg 2 tablets twice daily for 85 days
  Interventions: Dietary Supplement: Prosta-OK® Neo or Prosta-OK® Neo-matched placebo
- Tamsulosin and Prosta-OK® Neo-matched placebo (Placebo Comparator): Tamsulosin 0.2mg once daily and Prosta-OK® Neo-matched placebo 707mg 2 tablets twice daily for 85 days
  Interventions: Dietary Supplement: Prosta-OK® Neo or Prosta-OK® Neo-matched placebo

INTERVENTIONS:
Dietary Supplement: Prosta-OK® Neo or Prosta-OK® Neo-matched placebo — the patient planed to receive Tamsulosin 0.2mg once daily is randomized to the experiment group or placebo group. After randomization, the patient received Tamsulosin therapy with Prosta-OK® Neo or Prosta-OK® Neo-matched placebo 707mg 2 tablets twice daily for 85 days.

SUMMARY:
The aim of the study is to uses Prosta-OK® Neo that contains herb extracts including lycopene, phellinus linteus, pomegranate, pumpkin seed, selenium and zinc that have been demonstrated with functions of inhibiting 5-alpha reductase, antioxidant, anti-inflammation and regulating the synthesis of nitric oxide to explore whether Prosta-OK® can help reduce symptoms and elevate the quality of life in patients with mild to severe non-neurogenic male lower urinary tract symptoms receiving Tamsulosin therapy.

DETAILED DESCRIPTION:
Lower urinary tract symptoms (LUTS) are kind of uncomfortable subjective feelings reported from patients and are divided into three groups, storage, voiding, and postmicturition symptoms. Many epidemiological studies have pointed out that the prevalence of LUTS among individuals aged at least 40 years in the United States, the United Kingdom, Sweden, China, Taiwan, and South Korea is up to 60%. LUTS may cause mental health disorders such as anxiety and depression and affect lifestyle that leads to a negative impact on the quality of life. In recent years, there have been numerous academic or clinical studies that assess the improvement of plant and herb extracts in LUTS.

Prosta-OK® Neo is mainly comprised of herb extracts, including lycopene, phellinus linteus, pomegranate, pumpkin seed, selenium and zinc that have been demonstrated with functions of inhibiting 5-alpha reductase, antioxidant, anti-inflammation and regulating the synthesis of nitric oxide.

The aim of the study is to explore whether take Prosta-OK® 2 tablets for 85 days compared with placebo group can help reduce symptoms and elevate the quality of life in patients with mild to severe non-neurogenic male LUTS receiving Tamsulosin therapy.

ELIGIBILITY:
Inclusion Criteria:

* male between the ages of 30 and 55 when signing the informed consent form
* the subject was diagnosed with mild to severe non-neurogenic lower urinary tract symptoms and planed to receive Tamsulosin therapy
* the sum of International Prostate Symptom Score (IPSS) on questions 1 to 7 was 10 points or higher
* the subject can take medication via oral or nasogastric tube confirmed with the function of absorption by the principal investigator or co-principal investigators
* the subject was willing to corporate study-related procedures and sign the informed consent form

Exclusion Criteria:

* post-void residual urine volume greater than 200 mL or peak of maximum urine flow rate less than 5 mL/s
* total serum prostate-specific antigen higher than 10 ng/mL
* bladder outlet obstruction caused by reasons other than benign prostatic hyperplasia
* lower urinary tract symptoms caused by neurological disease such as Cerebrovascular Diseases, Parkinson's, dementia, Multiple Sclerosis (MS), spinal cord injuries (SCI), cauda equina syndrome, and Peripheral Neuropathy
* history or evidence of prostate cancer, male reproductive cancers, bladder cancer, and cancer of the ureter and urethra
* history or evidence of acute urinary retention (AUR)
* history or evidence of acute orthostatic hypotension
* with the urinary catheter or intermittent catheter
* stone in the urinary system
* Interstitial cystitis (IC), neurogenic bladder, overactive bladder (OAB) and Inflammatory Bowel Disease (IBD) within 3 mo prior to study entry
* chemotherapy or radiation therapy within 3 mo prior to study entry
* immunosuppressive therapy within 2 mo prior to study entry
* pelvic surgery or urinary surgery within 2 mo prior to study entry
* 5-alpha-reductase inhibitors use within 6 mo prior to entry or alpha-1-adrenergic blockers use within 2 w prior to entry
* the subject plans to use medication other than Tamsulosin such as alpha-blocker, 5-alpha-reductase inhibitors, antimuscarinic drugs, phosphodiesterase type 5 inhibitor (PDE5 inhibitors), Beta-3 agonists, desmopressin, diuretics, phenazopyridine, other drugs or foods are known to interact with tamsulosin and steroid or a nonsteroidal anti-inflammatory drug during participating in the study.
* the subject plans to receive cataract surgery during participating in the study or 1 mo after participating in the study.
* the subject took other therapies such as acupuncture or phytotherapy, including Saw Palmetto, Pygeum Africanum, Hypoxis Rooperi, Rye-pollen extract, and Pumpkin Seed extract within 2 w prior to entry.
* the subject took Chinese herbs such as Soaring Dragon Decoction, Rehmannia Right Formula, Powder for Five Types of Painful Urinary Dysfunction, Minor Bupleurum Decoction, Artemisiae Scopariae Decoction, Decoction to Enrich Yin and Direct Fire Downward, Tonifies Qi、Coptis Decoction to Relieve Toxicity and related modifications, Radix Rehmanniae, Cortex Moutan, Radix Pulsatillae, Herba Taraxaci, Herba Portulacae, Fructus Forsythiae, Flos Lonicerae, Herba Lophatheri, Fructus Gardeniae, Phellinus linteus within 7 days prior to entry.
* have a history of allergy to the ingredients of investigational product
* Serum Glutamic-Oxaloacetic Transaminase and serum Glutamic-Pyruvic Transaminase were more than three times of normal range or Serum creatinine less than 1.5 mg/dL
* have a history of substance abuse within 2 yr prior to entry
* participating in any clinical trial such as health food, herbal extracts, and drug within 30 days prior to entry
* have other significant diseases and confirmed by the principal investigator as non-eligible to be enrolled in the study

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-04 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
change in International Prostate Symptom Score from baseline on the sum of 1 to 7 questions | day 1 (before receiving therapy) and day 85
  compare the change in International Prostate Symptom Score from baseline between the experiment group and placebo group on the sum of 1 to 7 questions that are related to voiding symptoms. Scores of 0 to 7, 8 to 19, and 20 to 35 signify mild, moderate, and severe symptoms, respectively.

SECONDARY OUTCOMES:
change in International Prostate Symptom Score on questions 1, 3, and 5 that are related to voiding symptoms, questions 2, 4, and 7 that are related to storage symptoms, and question 8 that is related to the quality of life from baseline | day 1 (before receiving therapy) and day 85
  compare the change in International Prostate Symptom Score on questions 1, 3, and 5 that are related to voiding symptoms, questions 2, 4, and 7 that are related to storage symptoms, and question 8 that is related to the quality of life from baseline between the experiment group and placebo group. A higher score is indicated more severe in symptoms.
change in International Prostate Symptom Score from baseline by visit on the sum of 1 to 7 questions that are related to voiding symptoms and question 8 that is related to the quality of life | day 1 (before receiving therapy), day 15, day 29, and day 85
  compare the change in International Prostate Symptom Score from baseline by visit between the experiment group and placebo group on the sum of 1 to 7 questions that are related to voiding symptoms and question 8 that is related to the quality of life. A higher score is indicated more severe in symptoms or dissatisfaction in the quality of life.
change in interleukin 6, interleukin 8, tumor necrosis factor-alpha and interleukin 1 beta levels in expressed prostatic secretion from baseline by visit | day 1 (before receiving therapy), day 15, day 29, and day 85
  compare the change in interleukin 6, interleukin 8, tumor necrosis factor-alpha and interleukin 1 beta levels in expressed prostatic secretion collected from urine after a prostate massage from baseline by visit between the experiment group and placebo group.
change in maximum urinary flow rate from baseline. | day 1 (before receiving therapy) and day 85
  compare change in maximum urinary flow rate from baseline between the experiment group and placebo group.
change in amount of post voiding residual urine from baseline. | day 1 (before receiving therapy) and day 85
  compare change in amount of post voiding residual urine from baseline between the experiment group and placebo group.
percentage of patients with adverse reaction | day 1 (after receiving therapy) to day 85
  adverse reactions caused by the investigational product will be documented and recorded for analysis.
correlation of lifestyle factors on the severity of non-neurogenic male lower urinary tract symptoms assessed by the International Prostate Symptom Score | screening visit to day 85
  Lifestyle factors are assessed by self-designed questionnaires. The severity of non-neurogenic male lower urinary tract symptoms is assessed by the International Prostate Symptom Score, consisting of 8 questions, of which 1 to 7 questions are for evaluating the symptoms of voiding and question 8 is for evaluating the quality of life. A higher score is indicated more severe in symptoms or dissatisfaction in the quality of life.
correlation of the other external factors on the severity of non-neurogenic male lower urinary tract symptoms assessed by the International Prostate Symptom Score | screening visit to day 85
  The other external factors are assessed by self-designed questionnaires. The severity of non-neurogenic male lower urinary tract symptoms is assessed by the International Prostate Symptom Score, consisting of 8 questions, of which 1 to 7 questions are for evaluating the symptoms of voiding and question 8 is for evaluating the quality of life. A higher score is indicated more severe in symptoms or dissatisfaction in the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Ru HO, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chiayi Chang Gung Memorial Hospital, Chiayi County, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided